CLINICAL TRIAL: NCT06277856
Title: The Effect of Peer Interaction on Breastfeeding Self-Efficacy of Primiparas Sharing the Same Room With Mothers With Successful Postpartum Breastfeeding Experience; Randomised Controlled Study
Brief Title: Peer Interaction of Primiparas Sharing a Room With Multiparas With Successful Breastfeeding Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, AYSUN EKŞİOĞLU, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Aysun Eksioglu; Ayse Akyar (Other: Ege University)
Record Dates: First submitted 2023-12-25; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mothers
Keywords: Breastfeeding; Peer; interaction; Education; Hospital based; room
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Masking Description: In order to eliminate selection bias in the study, "block randomisation" method, one of the fixed probability randomisation methods, will be used and women who meet the inclusion criteria will be distributed to the intervention and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peer interaction (Experimental): The rooms will be arranged for two people and experienced and inexperienced mothers will be accommodated together. At a time when the mothers are available, the researcher will visit the mothers in their rooms, explain the purpose of the study and start the peer interaction session. In providing peer interaction, firstly, introductions will be made and the general condition of mothers and babies will be evaluated. The researcher will assess the breastfeeding status of the mothers and provide training on breastfeeding and breastfeeding.
  Interventions: Behavioral: Peer interaction/control
- control group (No Intervention): Women in this group benefit from all routine postnatal care services of the hospital. Each mother is guided to breastfeeding by the breastfeeding counsellor and receives training. This group will also be given a brochure by the researcher, their breastfeeding status will be evaluated and if they have any questions, they will be answered.

INTERVENTIONS:
Behavioral: Peer interaction/control — This study was planned as a randomised controlled study with a two-group pretest and posttest design.
  Arms: peer interaction

SUMMARY:
The World Health Organization (WHO) states that peer support breastfeeding education programs are effective interventions for improving breastfeeding outcomes. In this context, the WHO's Global Strategy for Infant and Young Child Feeding recommends the implementation of "lay health worker peer counselors" and "mother-to-mother support groups" to promote and support breastfeeding. The tenth step of the Baby-Friendly Hospital Initiative also emphasizes the importance of mother-to-mother support as a successful intervention for breastfeeding. However, in our country, there have been limited studies and efforts to provide peer education and support for breastfeeding. Although various valuable studies using different educational techniques have been conducted to improve breastfeeding rates, the integration of these programs into routine clinical practice remains insufficient. This study aims to implement a peer interactive education program in postpartum rooms to bring experienced and inexperienced mothers together, as part of the hospital routine. The project will focus on the development and implementation of a peer interactive education program and will investigate its impact on the breastfeeding self-efficacy of primiparous mothers. The research follows a two-group pre-test and post-test design, is non-blind, and uses randomized controlled methodology. Initially, the hospital rooms will be rearranged to accommodate the implementation of the peer support breastfeeding education module. Researcher midwives will provide a brief training to experienced peer educator mothers who have previously breastfed.Afterwards, the peer education program will be conducted when the experienced mother and primiparous mother are together in the room. The study emphasizes improving early postpartum breastfeeding success and aims to make peer interaction a routine part of hospital practice. The feasibility of implementing peer education in hospitals will be evaluated, considering its simplicity and practicality. The impact of peer interactions on the mother's breastfeeding self-efficacy and attitudes towards breastfeeding will be assessed.

Overall, this research aims to improve breastfeeding rates by implementing peer support programs in hospital settings and evaluating the outcomes of peer interactions in terms of the mother's breastfeeding self-efficacy and attitudes towards breastfeeding.

DETAILED DESCRIPTION:
Study Design: This project was planned as a two-group, non-blinded randomised controlled trial.

Ethical approval was obtained from the Medical Research Ethics Committee of a university for the conduct of the study (Date: 08.11.2022, Decision no: 22-11T/25).

Population and Sample of the Study: Mothers who were hospitalised in Izmir Democracy University Buca Seyfi Demirsoy Training and Research Hospital obstetrics and gynaecology ward, who met the inclusion criteria and volunteered to participate in the study will constitute the population of the study. A priori power analysis was performed using G.Power 3.1.9.2 package programme to determine the sample size. In the calculation made, with the assumption of 0.5 effect value for 80% power at 95% confidence interval, it was calculated as 128 women, 64 for the group in which peer supported breastfeeding education will be applied and 64 for the group in which standard education will be applied. In order to ensure homogeneity between the groups and to eliminate selection bias, the "block randomisation" method, one of the fixed probability randomisation methods, will be used in the study and women who meet the inclusion criteria will be distributed to the intervention and control groups.

Hypotheses of the study

1. H1: Breastfeeding self-efficacy of mothers who receive peer interaction after birth will be higher than the control group.
2. H1: The level of exclusive breastfeeding of mothers receiving peer interaction will be higher than that of mothers in the control group.

ELIGIBILITY:
Mothers to provide peer support

* Multipar
* Mothers with successful breastfeeding experience (Exclusive breastfeeding of the previous baby for at least 6 months, continued breastfeeding at the age of 2 years or older)
* At least secondary education graduate
* Singleton birth
* Vaginal birth (due to rapid mobilisation after birth and quicker adaptation to daily activities)
* with a child aged 5 years and under (limit for the age of the previous child for the memory factor regarding breastfeeding experience)
* Breastfeeding self-efficacy scale score of 60 and above (out of a total score of 70)
* No known or diagnosed psychiatric health problem in medical history
* Women without any health problem that may prevent breastfeeding will be included.

Intervention-Control group mothers

* Primipar
* 18 years and over
* Singleton birth
* No known or diagnosed psychiatric health problem in medical history
* Women who do not have any health problems that may prevent breastfeeding will be included.

Baby

* Born between 37-42 weeks
* Birth weight ≥2.5 kg and ≤3.9 kg
* 1 and 5 minute Apgar scores ≥8
* Not referred to neonatal intensive care unit

Exclusion criteria for individuals/patients in the study:

* Under 18 years of age
* Non-literate in Turkish
* Has a psychiatrically diagnosed health problem
* Developing a health problem that may prevent breastfeeding
* Taking medication that may jeopardise breastfeeding
* Women who do not want to participate will not be included in the study.

Exclusion criteria

* Requesting a room change
* Not wanting to/wanting to stop peer interaction within the scope of the room arrangement
* After settling in the room, those who did not want to answer the data collection tools for any reason/left the data collection tools unfinished
* Mothers who could not be reached in the postnatal 1st month follow-up will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
breastfeeding self-efficacy | After the participant is admitted to the labour ward, the first application within 1 hour (before the peer support intervention); At the 24th hour after the peer support module; It will be applied 3 times in the 1st postpartum month.
  It will be evaluated using the Breastfeeding Self-Efficacy Scale-SF. The scale consists of a total of 14 items and is 5-point Likert type. The lowest score that can be obtained from the scale is 14 and the highest score is 70; it is stated that breastfeeding self-efficacy increases in mothers with high scores.
exclusive breastfeeding rate | After the participant is admitted to the labour ward, the first application within 1 hour (before the peer support intervention); At the 24th hour after the peer support module; It will be applied 3 times in the 1st postpartum month.
  Exclusive breastfeeding is a physiological parameter. It will be evaluated according to the World Health Organisation classification system. Those who are exclusively breastfed, excluding ORS, drops, vitamins, minerals and medication will be grouped as "exclusively breastfed".

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Eksioglu, Assoc Prof, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed, the study protocol and data can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the work is completed
Access Criteria: not yet identified